CLINICAL TRIAL: NCT04562935
Title: Long-term Consequences of Admission for Pediatric Intensive Care Before One Year of Age
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gorm Greisen, consultant neonatologist, professor, Rigshospitalet, Denmark
Other Study IDs: VD-2019-47
Record Dates: First submitted 2020-09-15; First posted 2020-09-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric intensive care: Children admitted to a pediatric intensive care unit before one year of age and admitted for to days or more and treated with mechanical ventilation and alive at follow
  Interventions: Other: admission to pediatric intensive care with mechanical ventilation

INTERVENTIONS:
Other: admission to pediatric intensive care with mechanical ventilation — admission to pediatric intensive care with mechanical ventilation

SUMMARY:
This study is a retrospective cohort study. The PICU children will include all surviving children who were admitted to the PICU of Copenhagen University Hospital between 1st of January 2002 and 31st of December 2016.

A link to a questionnaire including the Strengths-and-Difficulties parental questionnaire evaluating neurodevelopmental- and behavioral impartment as well as question on current impairments and health, will be sent to parents. For the children aged between 11 and 17 years an additional self-rated questionnaire will be provided.

DETAILED DESCRIPTION:
This study is a retrospective cohort study. The PICU children will include all surviving children who were admitted to the pediatric intensive care section of the Department of Neonatology of Copenhagen University Hospital between 1st of January 2002 and 31st of December 2016.

The Strengths-and-Difficulties parental questionnaire evaluating neurodevelopmental- and behavioral impartment is web-based an hosted on a safe hospital server. The link will be sent to the universat digital post-box that all Danish citizens use for contact to the public authorities. For the children aged between 11 and 17 years an additional self-rated questionnaire will be provided. Furthermore, parents will answer questions on chronic illness, motor and sensory handicap, and special pedagogical support in day care institutions and school.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the PICU of Copenhagen University Hospital between 1st January 2002 to 31st of December 2016
* Age of admission > 28 days, if born > 37 + 0 or have reached the gestational age of > 40 weeks if the child is premature.
* Needing ≥ 2 days ventilator support during the PICU stay
* Valid civil registration number

Exlusion criteria:

- Death before follow-up

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Total difficulty score of the SDQ questionnaire | 2 to 18 years of age
  Total difficulty score of the Strengths and Difficulties Questionnaire

SECONDARY OUTCOMES:
Rate of cerebral palsy | 2 to 18 years of age
  cerebral palsy defined as 2 or higher on the GMFCS-scale

OTHER OUTCOMES:
Rate of learning disability | 2 to 18 years of age
  any educational or pedagogical support as reported by parents, more than 9 hours per week
Rate of chronic disease | 2-18 years
  any disease requiring continued medication and/or medical check-ups
Rate of visual impairment | 2-18 years
  that cannot be corrected by glasses or blind
Rate of hearing impairment | 2-18 years
  requiring amplification by hearing aid or deaf

CONTACTS AND LOCATIONS:
Overall Officials: gorm greisen, prof, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Gorm Greisen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Complex personal data, that cannot meaningfully be reduced to a level that will make re-identification possible